CLINICAL TRIAL: NCT01643590
Title: A Phase II Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of a Single Dose of JVS-100 Administered by Endomyocardial Injection to Cohorts of Adults With Ischemic Heart Failure
Brief Title: Study to Evaluate the Safety and Efficacy of JVS-100 Administered to Adults With Ischemic Heart Failure.
Acronym: STOP-HF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Juventas Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JTCS-004
Record Dates: First submitted 2012-07-10; First posted 2012-07-18 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Ischemic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo Injection
- 15 mg dose of JVS-100 (Experimental): 15 mg dose of JVS-100
  Interventions: Biological: JVS-100 15 mg dose Injection
- 30 mg dose of JVS-100 (Experimental): 30 mg dose of JVS-100
  Interventions: Biological: JVS-100 30 mg dose injection

INTERVENTIONS:
Biological: JVS-100 15 mg dose Injection — Intramyocardial Injection
  Arms: 15 mg dose of JVS-100
Biological: Placebo Injection — Intramyocardial Injection
  Arms: Placebo
Biological: JVS-100 30 mg dose injection — Intramyocardial Injection
  Arms: 30 mg dose of JVS-100

SUMMARY:
This is a randomized, double-blind, placebo controlled Phase II study is designed to assess the safety and efficacy of using JVS-100 to treat heart failure.

DETAILED DESCRIPTION:
90 subjects with ischemic cardiomyopathy will be randomized to receive a single dose of 15 or 30 mg of JVS-100 or matching placebo. Subjects will be randomized 1:1:1 to receive either placebo, 15 mg or 30 mg of JVS-100. Subjects will be monitored overnight for 18-24 hours post dose and have scheduled visits at 3 days post-injection for safety evaluations. All subjects will be scheduled for follow-up visits at approximately 30 days (1 month), 120 days (4 months), and 360 days (12 months) to assess safety and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign informed consent
* Greater than or equal to 18 years of age
* Subjects with impaired 6 minute hall walk distance
* Impaired quality of life as measured by Minnesota LWHF questionnaire
* Ischemic cardiomyopathy without an acute coronary syndrome within the last 6 months
* Residual well-demarcated region of LV systolic dysfunction defined as at least 3 consecutive segments of abnormal wall motion by echocardiography read at the echocardiography core laboratory
* LVEF ≤40% measured by echocardiography read at the echocardiography core laboratory
* Must meet wall thickness criteria
* Subject has an implanted, functional AICD
* Subjects with diabetes must have had an ophthalmologist exam within the last year showing no active proliferative retinopathy
* Subject receiving stable optimal pharmacological therapy defined as:

  * ACE inhibitor and/or ARB, and Beta-blocker for 90 days with stable dose for 30 days unless contraindicated
  * Diuretic in subjects with evidence of fluid retention
  * ASA unless contraindicated
  * Statin unless contraindicated
  * Aldosterone antagonist per physician discretion

Exclusion Criteria:

* Planned revascularization within 30 days following enrollment
* Estimated Glomerular Filtration Rate < 30 ml/min*
* Signs of acute heart failure within 24 hours of scheduled injection
* History of aortic valve regurgitation classified as "moderate" or severe
* Moderate/Severe aortic stenosis defined as AVA <1.5 cm2

Note: Patient should not be excluded if the patient's medical records document that within the last 6 months the patient has either:

* no aortic stenosis
* mild aortic stenosis
* normal aortic valve
* normal aortic pressure gradient
* aortic pressure gradient < 20 mmHg

  * Presence of an artificial aortic valve
  * Subjects with aortic aneurysm >3.8 cm
  * Mitral regurgitation defined as "severe" measured by echocardiography at the clinical site.
  * Patients with planned mitral valve repair or replacement surgery
  * Any patient with a history of cancer will be excluded unless:
* The cancer was limited to curable non-melanoma skin malignancies and/or
* The cancer was removed by a successful tumor resection, with or without radiation or chemotherapy treatment, 5 years or more prior to enrollment in this study without recurrence

Subjects must have the following results on age appropriate cancer screenings:

* Subjects age 50 or older have had a Fecal occult blood test (FOBT) or fecal immunochemical test (FIT) that was negative within the last year
* Women age 30 or older have had a PAP test that was negative within the last 3 years
* Women age 40 or older have had a mammogram that was negative within the last year
* Men above age 45 have had a Prostate-Specific Antigen (PSA) blood test and digital rectal examination (DRE) that was negative within the last year
* At the request of the site principal investigator, any subject with a non-negative result thought to be due to a non-cancer-related condition will be evaluated by the medical monitor for enrollment

Exclusion Criteria (ctd):

* Subjects with persistent or chronic atrial fibrillation will be excluded unless:

  * A stable, regular heart rate is maintained with a biventricular pacemaker
  * A stable, regular heart rate is maintained with a univentricular pacemaker pacing less than or equal to 40% of the time
* Subjects with Biventricular pacing device implant within the last 3 months OR previously implanted Biventricular pacing device with programming planned to be reoptimized following enrollment in this trial
* Previous solid organ transplant
* Subjects with greater than 40% univentricular RV Pacing
* Subjects with uncontrolled diabetes defined as HbA1c >9.0%
* Inability to complete 6 minute walk or treadmill exercise test
* Participation in an experimental clinical trial within 30 days prior to enrollment
* Any subject who has been enrolled in a gene or stem cell therapy cardiac trial within the last year
* Life expectancy of less than 1 year
* Positive pregnancy test (serum βHCG) in women of childbearing potential and/or unwillingness to use contraceptives or limit sexual activity as described in Section 8.2.1 below
* Unwillingness of men capable of fathering a child to agree to use barrier contraception or limit sexual activity as described in Section 8.2.1 below
* Subjects who are breast feeding
* Subjects with a positive test results for hepatitis B/C and/or HIV
* Total Serum Bilirubin >4.0 mg/dl
* Aspartate aminotransferase (AST) > 120 IU/L
* Alanine aminotransferase (ALT) > 135 IU/L
* Alkaline phosphatase (ALP) >300 IU/L
* Clinically significant elevations in PT or PTT relative to laboratory norms
* Any subject with a known existing LV thrombus or has an LV thrombus detected during the screening period of this study.
* Subjects with Rutherford class 5 or 6 critical limb ischemia
* Subject with severe chronic obstructive pulmonary disease (COPD)
* Any subject requiring home oxygen use
* Subjects with a history of Systemic Lupus Erythematosus (SLE) flare
* History of drug or alcohol abuse within the last year
* A subject will be excluded if he/she is unfit for the trial based on the discretion of the site Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Impact of JVS-100 injection on Six Minute Walk Distance (6MWD) at 4 month follow-up | 4 Months
  To investigate the impact of single doses of JVS-100 (either 15 or 30 mg) delivered via endomyocardial injection through the BioCardia Helical Infusion catheter on 6 minute walk distance compared to placebo at 4 months post-dosing
Impact of JVS-100 injection on Quality of Life at 4 month follow-up | 4 months
  To investigate the impact of single doses of JVS-100 (either 15 or 30 mg) delivered via endomyocardial injection through the BioCardia Helical Infusion catheter on quality of life measured by the Minnesota Living with Heart Failure Questionnaire compared to placebo at 4 months post-dosing

SECONDARY OUTCOMES:
Impact of JVS-100 Injection on Quality of Life | 12 Months
  To investigate the impact of single doses of JVS-100 (either 15 or 30 mg) delivered via endomyocardial injection through the BioCardia Helical Infusion catheter on quality of life measured by the Minnesota Living with Heart Failure Questionnaire compared to placebo at 12 months post-dosing
Impact of JVS-100 Injection on NYHA class | 4 months
  To investigate the impact of single doses of JVS-100 (either 15 or 30 mg) delivered via endomyocardial injection through the BioCardia Helical Infusion catheter on NYHA class compared to placebo at 4 months post-dosing
Impact of JVS-100 Injection on LVEF | 4 months
  To investigate the impact of single doses of JVS-100 (either 15 or 30 mg) delivered via endomyocardial injection through the BioCardia Helical Infusion catheter on Left Ventricular Ejection Fraction as measured by echocardiography compared to placebo at 4 months post-dosing
Impact of JVS-100 Injection on Time to First Heart Failure Decompensation | Up to 12 months
  To investigate the impact of single doses of JVS-100 (either 15 or 30 mg) delivered via endomyocardial injection through the BioCardia Helical Infusion catheter on the time to first heart failure decompensation compared to placebo
Impact of JVS-100 Injection on Major Adverse Cardiac Events | Up to 12 months
  To investigate the impact of single doses of JVS-100 (either 15 or 30 mg) delivered via endomyocardial injection through the BioCardia Helical Infusion catheter on the number of major adverse cardiac events (MACE) compared to placebo
Impact of JVS-100 Injection on number of adverse events | Up to 12 months
  To investigate the impact of single doses of JVS-100 (either 15 or 30 mg) delivered via endomyocardial injection through the BioCardia Helical Infusion catheter on the number of adverse events compared to placebo
Impact of JVS-100 Injection on number of serious adverse events | Up to 12 months
  To investigate the impact of single doses of JVS-100 (either 15 or 30 mg) delivered via endomyocardial injection through the BioCardia Helical Infusion catheter on the number of serious adverse events compared to placebo

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Cardiology PC, Birmingham, Alabama
  - University of Florida, Gainesville, Florida
  - Pepin Heart Institute, Tampa, Florida
  - Iowa Heart Center, Des Moines, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Spectrum Health, Grand Rapids, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - Summa Health System, Akron, Ohio
  - The Lindner Center at the Christ Hospital, Cincinnati, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Baylor Healthcare, Dallas, Texas
  - University of Utah, Salt Lake City, Utah